CLINICAL TRIAL: NCT04628988
Title: A Phase 1, Open-label, Functional Imaging Study to Assess Whether CC-90011 Reverses the Castration Resistance Due to Lineage Switch in Subjects With Metastatic Castration-resistant Prostate Cancer (mCRPC) Who Have Failed Enzalutamide as Last Prior Therapy, Followed by a Dose Finding Study of CC-90011 Combined With Abiraterone and Prednisone
Brief Title: A Study of CC-90011 and Comparators in Participants With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-90011-PCA-001; U1111-1257-9342 (Registry Identifier: WHO)
Record Dates: First submitted 2020-10-27; First posted 2020-11-16 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Prostatic Neoplasms
Keywords: mCRPC; AR; enzalutamide; abiraterone; LSD1; Prostate Cancer; CC-90011; Prednisone
MeSH Terms: conditions — Prostatic Neoplasms | interventions — pulrodemstat besilate; abiraterone; Abiraterone Acetate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CC-90011 in combination with Abiraterone and Prednisone (Experimental): Oral administration (PO) of CC-90011 monotherapy administered once per week (QW), for 4 weeks. From cycle 2 onwards, all participants will receive 60 mg of CC-90011 PO QW, in combination with 100 mg of abiraterone PO daily, and 5 mg of prednisone PO every 12 hours (10mg QD)
  Interventions: Drug: CC-90011; Drug: Abiraterone; Drug: Prednisone

INTERVENTIONS:
Drug: CC-90011 — Capsule
Drug: Abiraterone — Tablet
  Other Names: Zytiga
Drug: Prednisone — Tablet
  Other Names: Deltasone

SUMMARY:
This is an open-label, positron emission tomography (PET) imaging Proof of Biology (POB) study to determine whether CC -90011 reverses, by the induction of androgen receptor (AR) expression, the castration resistance, due to lineage switch, in participants with mCRPC that have failed enzalutamide as last prior therapy. This study aims to assess whether CC-90011 can induce AR expression and, consequently, re-sensitize tumors to anti-hormonal therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is a male ≥ 18 years of age the time of signing the informed consent form (ICF).
2. Histologically confirmed adenocarcinoma of the prostate.
3. Surgically or medically castrated, with testosterone levels of < 50 ng/dL (<2.0 nM). If the participant is being treated with luteinizing hormone-releasing hormone (LHRH) agonists/antagonists (participant who have not undergone orchiectomy) this therapy must have been initiated at least 4 weeks prior to Cycle 1 Day 1 and must be continued throughout the study.

   Participants must have failed prior therapy with enzalutamide or apalutamide
   * Has completed at least 12 weeks of prior continuous therapy with enzalutamide or apalutamide .
   * Has been without enzalutamide, or apalutamide treatment for >30 days prior to initiation of study treatment.
4. Documented prostate cancer progression as assessed by the investigator with one of the following:

   * Prostate-specific antigen (PSA) progression defined by a minimum of 3 rising PSA levels with an interval of ≥1 week between each determination. The PSA value at screening must be ≥1 µg/L (1 ng/mL) if PSA is the only indication of progression; participants on systemic glucorticoids for control of symptoms must have documented PSA progression by PCWG3 criteria while on systemic glucocorticoids prior to commencing Cycle 1 Day 1 treatment.
   * Radiographic progression of soft tissue disease by RECIST 1.1 or bone metastasis with 2 or more documented new bone lesions on a bone scan with or without PSA progression.
5. Participants must have FDHT lesion >2 cm lesion that has an SUVmax of 2.9 or less in bone, or 2.4 or less in soft tissue, or two or more smaller lesions that meet those criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at Screening.
7. Participants must have the following laboratory values:

   * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L without growth factor support for 7 days (14 days if participant received pegfilgastrim)
   * Hemoglobin (Hgb) ≥ 9 g/dL (≥ 90 g/L or > 5.59 mmol/L)
   * Platelet count (plt) ≥ 100 x 109/L
   * Serum potassium concentration within normal range, or correctable with supplements
   * Serum AST/SGOT and ALT/SGPT ≤ 3.0 x Upper Limit of Normal (ULN) or ≤ 5.0 x ULN if liver metastases are present
   * Serum total bilirubin ≤ 1.5 x ULN (≤ 2 x ULN in case of documentened Gilbert).
   * Participants must have serum albumin ≥ 3.0 g/dL
   * Serum creatinine ≤ 1.5 x ULN, or measured glomerular filtration rate (GFR) ≥ 60 mL/min/1.73m2 using an exogenous filtration marker such as iohexol, inulin, 51Cr EDTA or 125I iothalamate. In cases where the serum creatinine is < 1,5xULN, there is no need to calculate GFR.
   * PT (or INR) and activated partial thromboplastin time (APTT)

     1. within normal range (Part A)
     2. ≤1.5 ULN

Exclusion Criteria:

1. Participant has received anti-cancer therapy (either approved or investigational) < 4 weeks or 5 half-lives, whichever is shorter, prior to Cycle 1 Day 1.

   - < 42 days for prior nitrosureas or mitomycin C
2. Toxicities resulting from prior systemic cancer therapies must have resolved to ≤ NCI CTCAE Grade 1 prior to starting CC-90011 treatment (with exception of Grade 2 peripheral neuropathy and alopecia).
3. Previous anaphylactic reaction to either FDHT or FDG.
4. Participant has undergone major surgery ≤ 4 weeks or minor surgery ≤ 2 weeks prior to Cycle 1 Day 1 or who have not recovered from surgery.
5. Participant has completed any radiation treatment < 4 weeks prior to Cycle 1 Day 1 or < 2 weeks for palliative bone radiotherapy (single fraction). Participants with > 25% of myelopoietic bone marrow radiation are not allowed to be enrolled on this study.
6. Participant has persistent diarrhea due to a malabsorptive syndrome (such as celiac sprue or inflammatory bowel disease) ≥ NCI CTCAE Grade 2, despite medical management), or any other significant GI disorder that could affect the absorption of CC-90011.
7. Participant with symptomatic or uncontrolled ulcers (gastric or duodenal), particularly those with a history of and/or risk of perforation and GI tract hemorrhages.
8. Participant with any hemorrhage/bleeding event > CTCAE Grade 2 or haemoptysis > 1 teaspoon within 4 weeks prior to the first dose
9. Symptomatic and untreated or unstable central nervous system (CNS) metastases or clinically significant spinal cord compression.

   * Participant recently treated with whole brain radiation or stereotactic radiosurgery for CNS metastases must have completed therapy at least 4 weeks prior to Cycle 1, Day 1 and have a follow-up brain computed tomography (CT) or magnetic resonance imaging (MRI) demonstrating either stable or improving metastases 4 or more weeks after completion of radiotherapy (the latter to be obtained as part of the Screening Assessments, refer to Section 6.1)
   * Participant must be asymptomatic and off steroids or on stable dose of steroids for at least 4 weeks (?10 mg/day prednisone equivalent)
10. Participant has known symptomatic acute or chronic pancreatitis.
11. Participant with severe hepatic impairment (Child-Pugh Class C).
12. Medical castration with LHRH analogue is not permitted at any time during treatment with abiraterone and prednisone if not started at least 4 weeks prior to Cycle 2 Day 1.
13. Participant has impaired cardiac function or clinically significant cardiac diseases, including any of the following considered to be clinically significant by the subject's physician:

    * LVEF < 45% as determined by multiple gated acquisition scan (MUGA) or echocardiogram (ECHO)
    * Complete left bundle branch or bifascicular block
    * Congenital long QT syndrome
    * Persistent or clinically meaningful ventricular arrhythmias or atrial fibrillation.
    * QTcF ≥ 450 msec on Screening ECG (mean of triplicate recordings)
    * Unstable angina pectoris or myocardial infarction ≤ 6 months prior to starting CC-90011
14. Participant has other clinically significant heart disease such as congestive heart failure requiring treatment or uncontrolled hypertension (blood pressure ? 160/95 mm Hg).
15. Participants who are known to be human immunodeficiency virus (HIV) positive with an acquired immunodeficiency syndrome (AIDS) defining opportunistic infection within the last year, a detectable viral load, or a current CD4 count < 350 cells/uL.
16. Participant has untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 500 IU/mL (2500 copies/mL), or active hepatitis C. Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B (HBV DNA < 500 IU/mL), and cured hepatitis C participants can be enrolled.
17. Participant with ongoing treatment with chronic, therapeutic dosing of anticoagulants (eg, warfarin, low molecular weight heparin, Factor Xa inhibitors, thrombin antagonist). Low dose low molecular weight heparin for catheter maintenance and for short-term prophylaxis for participants with prior pulmonary embolism (PE) and deep vein thrombosis (DVT) are permitted under careful consideration by the Investigator.
18. Participant has a history of concurrent second cancers requiring active, ongoing systemic treatment.
19. Participant has any significant medical condition (eg, active or uncontrolled infection or renal disease), the presence of laboratory abnormalities, or psychiatric illness that would prevent the participant from participating (or compromise compliance) in the study or would place the participant at unacceptable risk if he/she were to participate in the study.
20. Participants with poor bone marrow reserve as assessed by Investigator such as in the following conditions of:

    * Having received extensive bone radiotherapy
    * Having experienced several episodes of bone marrow aplasia in previous treatments
    * Requiring regular hematopoietic support (blood transfusion, erythropoietin, GCSF)
21. Participant has any condition that confounds the ability to interpret data from the study.
22. Participant does not tolerate the study drug components.
23. Previous SARS-CoV-2 infection within 10 days for mild or asymptomatic infections or 20 days for severe/critical illness prior to Cycle 1 Day 1 (C1D1).

    • Acute symptoms must have resolved and based on investigator assessment in consultation with the Study Sponsor Physician, there are no sequelae that would place the subject at a higher risk of receiving study treatment
24. Previous SARS-CoV-2 vaccine within 7 days of C1D1. For vaccines requiring more than one dose, the full series (e.g. both doses of a two-dose series) should be completed prior to C1D1 when feasible and when a delay in C1D1 would not put the study subject at risk.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2021-07-28 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Assessment of androgen receptor (AR) level | From Screening to the end of cycle 3 (each cycle is 28 days)
  FDG/FDHT PET imaging will be compared with Screening to Cycle 1 (each cycle is 28 days) and from Cycle 1 to Cycle 3 (Cycle 2-3 is combined therapy period) to assess changes in AR expression.

SECONDARY OUTCOMES:
Safety and tolerability assessed by Adverse events (AEs) | From the time the subject signs the ICF until 90 days (± 3 days) after the last dose of study medication
  All AEs will be monitored and recorded from the time the subject signs the ICF until 90 days (± 3 days) after the last dose of study medication. For SAEs made known to the Investigator at any time thereafter that are suspected of being related to study drug, must be reported. For subjects who have high blood pressure related to abiraterone treatment, blood pressure monitoring every 2 weeks should continue after discontinuation of abiraterone until the blood pressure normalizes or returns to pre-enrollment levels.
Safety and tolerability assessed by dose-limiting toxicities (DLTs) | Through study completion, Up to 1.5 years
  DLTs will be assessed using the NCI CTCAE criteria, version 5.0. An event will be considered a DLT if the event is attributed (definitely, probably or possibly) to study treatment during Cycle 2 (4weeks) consistent with CC-90011 in combination with abiraterone and prednisone
Assessment of anti-tumor activity | Through study completion, Up to 3 years
  Anti-tumor activity will be assessed based on Prostate Cancer Clinical Trials Working Group (PCWG3) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 101, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com